CLINICAL TRIAL: NCT06929884
Title: Effectiveness, Safety, and Economic Evaluation of Goserelin Microspheres for Injection and Goserelin Sustained-Release Implants in Prostate Cancer Patients: A Real-World Study
Status: Active, not recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Rui Yang, Associate professor of pharmacy, Qianfoshan Hospital
Other Study IDs: LCYX-YR-20230103
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancers
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Patients receiving 3.6 mg goserelin sustained-release implants (subcutaneous).
- Intervention:: Patients receiving 3.6 mg goserelin microspheres (intramuscular).

SUMMARY:
Prostate cancer (PC) is the most common malignancy in the male genitourinary system. In China, both the incidence and mortality rates of PC have shown a significant upward trend in recent years. Chinese patients are typically diagnosed at older ages with higher preoperative prostate-specific antigen (PSA) levels compared to Western populations, indicating a more aggressive disease phenotype. This may explain the lower 5-year survival rates in Chinese PC patients. Over the past three decades, the age-standardized incidence of PC in China has surged by 95.2%, while the global rate increased by only 13.2%. Conversely, global PC mortality decreased by 15.7%, whereas China saw a mere 5.3% reduction. The high economic burden on patients and healthcare systems underscores the urgency of optimizing treatment strategies. Direct annual medical costs for PC in China average $3,500 per patient, with drug expenses accounting for over 60% and out-of-pocket payments comprising approximately 20%. These costs far exceed those of other malignancies, posing sustainability challenges for families and insurance systems. Androgen deprivation therapy (ADT), including surgical or chemical castration, remains the cornerstone for advanced PC. Chemical castration via luteinizing hormone-releasing hormone (LHRH) agonists or antagonists offers comparable survival benefits to surgical castration but with improved quality of life. Goserelin, a synthetic GnRH analog, has been widely used since 1987. Current formulations include a sustained-release implant (10.8 mg/3.6 mg) administered subcutaneously every 28 days using a 16G needle (outer diameter: 1.6 mm), which may cause injection-site injuries, and a newer microsphere formulation (3.6 mg) delivered intramuscularly via a 21G needle (outer diameter: 0.8 mm), enhancing patient tolerance. While Phase III trials showed no significant efficacy differences between the two formulations, real-world evidence is lacking. This retrospective cohort study aims to evaluate the effectiveness, safety, and cost-effectiveness of both formulations using real-world data.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients with histologically confirmed prostate cancer (PC) deemed suitable for endocrine therapy (excluding neoadjuvant endocrine therapy).

2. At least 18 years old 3. Prescribed 3.6 mg goserelin every 4 weeks as monotherapy or in combination with anti-androgen therapy.

Exclusion Criteria:

* 1. Hypersensitivity to LHRH, its analogs, or any component of goserelin. 2. Previous or concurrent hormone therapy, except for conventional anti-androgen therapy administered within 2 weeks before goserelin treatment.

  3. Diagnosis or suspicion of hormone-resistant PC, history of hypophysectomy, adrenalectomy, or pituitary lesions.

  4.Scheduled for radical radiotherapy (adjuvant radiotherapy post-radical prostatectomy [RP] combined with goserelin is permitted) or planned neoadjuvant hormone therapy prior to RP.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Hospitalized male patients diagnosed with PC between 2020 and 2025 at Shandong First Medical University Affiliated Hospital (Qianfoshan Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Serum testosterone | baseline, 1, 6, 12, and >12 months
  Serum testosterone
PSA levels | baseline, 1, 6, 12, and >12 months
percentage of patients achieving testosterone suppression (≤50 ng/dL and ≤20 ng/dL) | baseline, 1, 6, 12, and >12 months
digital rectal examination (DRE) | baseline, 1, 6, 12, and >12 months

SECONDARY OUTCOMES:
Imaging results (bone scans, pelvic/abdominal imaging), treatment adherence, adverse events (injection-site reactions), metabolic changes, hepatic/renal dysfunction), and cost-effectiveness analysis (CEA). | >12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China